CLINICAL TRIAL: NCT06882356
Title: The Glaucoma and Retinopathy Screening Study (GRaSS)
Brief Title: The Glaucoma and Retinopathy Screening Study
Acronym: GRaSS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts Eye and Ear Infirmary (Other)
Collaborators: Centers for Disease Control and Prevention (U.S. Federal Agency)
Responsible Party: Principal Investigator, David Steven Friedman, Professor of Ophthalmology, Massachusetts Eye and Ear Infirmary
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: 2024p003709
Record Dates: First submitted 2025-03-10; First posted 2025-03-18 (Actual); Last update posted 2025-08-28 (Actual); Status verified 2025-06

CONDITIONS: Glaucoma
MeSH Terms: conditions — Glaucoma

STUDY DESIGN:
Intervention Model Description: This study uses a prospective interventional model to evaluate the effectiveness of integrating AI-based glaucoma screening with existing diabetic eye disease (DED) screening among diabetic patients. Participants will have fundus images assessed by AI for glaucoma in addition to DED, and have intraocular pressure measurement measured. Suspected glaucoma cases will receive virtual perimetry testing for confirmation, and those diagnosed with glaucoma will be referred for follow-up care. This study aims to compare glaucoma detection rates between combined DED and glaucoma screening versus DED-only screening, ultimately supporting early glaucoma detection and enhancing care access in underserved communities.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Combined DED and Glaucoma Screening (Experimental): Participants in this arm will have fundus photographs that are taken as a part of standard clinical care analyzed by AI for signs of glaucoma in addition to for diabetic retinopathy. They will also have intraocular pressure measured. If the AI detects possible glaucoma, participants will undergo virtual perimetry testing for further assessment.
  Interventions: Device: AI-based glaucoma screening; Device: IOP measurement; Device: Virtual Reality Visual Field Testing
- DED Screening Only (Control Arm) (No Intervention): Participants in this arm will undergo diabetic eye disease (DED) screening only for routine clinical care. This includes fundus photography for AI assessment of signs of diabetic retinopathy.

INTERVENTIONS:
Device: AI-based glaucoma screening — AI analysis of fundus photographs to detect signs of glaucoma, added to AI-based diabetic eye disease screening performed for routine clinical care
  Arms: Combined DED and Glaucoma Screening
Device: IOP measurement — Intraocular pressure measurement by Icare tonometer
  Arms: Combined DED and Glaucoma Screening
Device: Virtual Reality Visual Field Testing — Virtual Reality Visual Field Testing by the Olleyes device for participants suspected of having glaucoma
  Arms: Combined DED and Glaucoma Screening

SUMMARY:
The goal of this clinical trial is to learn if a new screening approach including an artificial intelligence algorithm that analyzes fundus photographs, measurement of eye pressure and visual field testing works to screen for glaucoma.

Participants will:

Have an image of their fundus (back of the eye) taken as part of their diabetic eye screening Have a measurement of their eye pressure If needed, have a test of their side vision using a headset

DETAILED DESCRIPTION:
Study Overview: This study is a prospective, interventional clinical trial designed to evaluate the effectiveness of an artificial intelligence (AI)-based screening program within community health settings. This study targets especially diabetic patients because they have higher risks of developing glaucoma. By integrating glaucoma screening into existing diabetic eye disease (DED) screenings, the study aims to identify cases of glaucoma earlier, thereby preventing or delaying progression to blindness.

Background: Glaucoma is a chronic eye disease that causes progressive optic nerve damage, often leading to irreversible vision loss. Early detection is critical, as glaucoma is typically asymptomatic in its early stages. Individuals with diabetes are at an elevated risk for glaucoma, making it crucial to develop accessible screening methods. Current DED screening programs already utilize fundus photography for diabetic retinopathy. Adding glaucoma screening to these existing DED screenings may provide an efficient and cost-effective solution to reach high-risk populations without requiring additional clinic visits.

Study Hypothesis: The hypothesis of this study is that incorporating AI-driven glaucoma screening into standard DED screenings will increase the detection rate of glaucoma in high-risk populations compared to DED screening alone. This combined approach is expected to yield better clinical outcomes by enabling early diagnosis and treatment while being cost-effective.

Expected Outcomes and Impact: This study is expected to provide valuable insights into the effectiveness of integrating AI-based glaucoma screening into existing screening programs for diabetic eye disease. If successful, this combined screening approach could be a cost-effective model for other community health settings, leading to earlier detection of glaucoma and improved patient outcomes. By making glaucoma screening more accessible the study aims to reduce health disparities and support preventive eye care.

ELIGIBILITY:
* Individuals with diabetes undergoing AI-based screening for diabetic retinopathy using the LumineticsCore (Digital Diagnostics) system for clinical care at primary care centers.
* Individuals who are able and willing to provide informed consent for participation in the study.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2000 (Estimated)
Dates: Start 2025-07-16 (Actual); Primary Completion 2030-09 (Estimated); Study Completion 2030-09 (Estimated)

PRIMARY OUTCOMES:
Glaucoma detection | 1 year from initial screening
  This primary outcome measure will assesses the proportion of participants who receive a glaucoma diagnosis in the combined DED and glaucoma screening group compared to the DED-only screening group. Glaucoma diagnosis in the intervention group is based on AI-assisted analysis of fundus photography, intraocular pressure, and virtual reality perimetry testing for confirmation.

SECONDARY OUTCOMES:
Cost-Effectiveness of Combined Screening vs. DED-Only Screening | 1 year from initial screening
Participant Satisfaction with Screening Process | Day of screening
  This measure assesses participant satisfaction with the glaucoma screening process. Satisfaction will be evaluated through a participant satisfaction survey.
Participant knowledge about glaucoma | Day of screening
  This measure assesses participants' knowledge about glaucoma. Knowledge will be assessed through a questionnaire (NEI Glaucoma Eye-Q test).

CONTACTS AND LOCATIONS:
Overall Officials: David S Friedman, MD, PhD, MPH, Principal Investigator — Massachusetts Eye and Ear
Locations (5):
- United States (5):
  - Brigham and Women's Primary Care Associates of Longwood, Boston, Massachusetts
  - MGH Chelsea HealthCare Center, Chelsea, Massachusetts
  - NSPG Lynn, Lynn, Massachusetts
  - NSPG Salem, Salem, Massachusetts
  - NSPG Saugus, Saugus, Massachusetts

IPD SHARING:
Plan to Share IPD: Yes
Deidentified study data
Time Frame: After study completion
Access Criteria: Data sharing will require adherence to Mass General Brigham institutional and IRB policies. External researchers will need to contact the Principal Investigator to request data and complete a Data Use Agreement. Only deidentified data will be shared.